CLINICAL TRIAL: NCT06226987
Title: Molecular Imaging in Fabry Disease of the Heart
Status: Recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Jason Tarkin, Wellcome Clinical Research Career Development Fellow & Honorary Consultant Cardiologist, University of Cambridge
Other Study IDs: A095007
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Fabry Disease, Cardiac Variant
MeSH Terms: conditions — Fabry Disease, Cardiac Variant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabry Disease with cardiac involvement
  Interventions: Diagnostic Test: 68Ga-DOTATATE PET/MRI

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTATATE PET/MRI — PET/MRI scanning

SUMMARY:
Better methods for early detection of cardiac involvement in Fabry disease are needed to inform clinical management decisions that can help prevent or slow the progression of cardiac complications. In the Molecular Imaging of Inflammation in Fabry Disease of the Heart study, the investigators will test the use of 68Ga-DOTATATE PET/MRI for identifying myocardial inflammation in patients with Fabry disease.

DETAILED DESCRIPTION:
Fabry disease (OMIM 30150) is caused by mutations in the gene (AGAL) encoding for the lysosomal enzyme α-galactosidase A. Diminished activity of this enzyme results in progressive accumulation of its substrate globotriaosylceramide (Gb3) in the lysosomes of various cell types, including vascular endothelial cells, cardiomyocytes, valvular fibrocytes, conduction cells. The involvement of the heart in Fabry disease results in rhythm disturbances, progressive hypertrophy and scarring of the left ventricle leading to diastolic and systolic dysfunction.

Conventional diagnostic methods such as electrocardiography, transthoracic echocardiography and even magnetic resonance imaging (MRI) are not sensitive enough to detect early damage to myocardial tissue in Fabry disease. Identifying subtle early changes, at a point when specific treatment may be optimized, is therefore an area of ongoing interest. Early perspectives on Fabry heart involvement concentrated on the left ventricular hypertrophy. Later the widespread use of Cardiac MRI introduced the role of fibrosis, as suggested by the appearance of late gadolinium enhancement (LGE) in characteristic areas of the myocardium. Most recently, detection of oedema by T2-weighted imaging and/or T2-mapping on MRI, as well as 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) scanning have pointed to the possibility of focal inflammation as a causative factor in progression of the myocardial disease to replacement fibrosis, with its attendant risk of fatal arrhythmia and cardiac decompensation. Whether the oedema signal on MRI sequences truly represents tissue inflammation in Fabry disease and whether LGE fully corresponds to replacement fibrosis remains unknown. Circulating markers of inflammation and immune activation are elevated in Fabry cardiomyopathy, but no fully specific marker has yet been found to correspond to either myocardial focal oedema or LGE.

Although MRI is important for diagnosis and risk stratification in patients with cardiac involvement in Fabry disease, findings such as LGE, myocardial oedema and native T1 mapping tell the clinician little that is specific about the underlying disease mechanisms. Moreover, early inflammatory changes may occur in Fabry disease before the manifestation of such abnormalities are detectable by MRI. By combining PET imaging of myocardial inflammation with detailed MRI assessments of cardiac function, structure and tissue characterisation, hybrid PET/MRI has the potential to offer a comprehensive non-invasive workup for patients with Fabry disease.

Previous work has shown that 68Ga-DOTA-(Tyr3)-octreotate (DOTATATE), a somatostatin receptor PET tracer used in oncology imaging, can be re-purposed to image inflammation in the cardiovascular system. This method could be of particular use in conditions associated with focal myocardial inflammation such as Fabry disease because of low physiological expression of somatostatin receptors in healthy heart muscle, and therefore low background PET signal. Here, the investigators will investigate the use of 68Ga-DOTATATE PET/MRI for identifying myocardial inflammation in patients with Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants >18 years old
* Able to give written, informed consent and to lie flat
* Have Fabry disease based on molecular diagnosis (at a minimum, documented enzyme deficiency in males and documented pathogenic mutation in females)
* Cardiac MRI within 3 years documenting cardiac involvement in Fabry disease (left ventricular hypertrophy and/or late gadolinium enhancement and/or myocardial oedema)

Exclusion Criteria:

* Any other diagnosis associated with cardiac muscle inflammation, including myocarditis
* Previous gene therapy
* Contra-indication to MRI scanning or intravenous gadolinium contrast (prior contrast reaction or chronic kidney disease with eGFR <30 mL/min/1.73 m2)
* Women of child bearing potential not using adequate contraception
* Uncontrolled atrial fibrillation
* Any medical condition, in the opinion of the investigator, that prevents the participant from lying flat during scanning, or from participating in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with cardiac involvement in Fabry disease assessed by MRI
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
PET imaging vs. oedema detected by MRI | Baseline
  Concordance between 68Ga-DOTATATE PET signal and myocardial oedema on MRI assessed by T2-weighted imaging
PET imaging vs. fibrosis detected by MRI | Baseline
  Concordance between 68Ga-DOTATATE PET signal and myocardial fibrosis detected by late gadolinium enhancement MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tarkin JM, Joshi FR, Evans NR, Chowdhury MM, Figg NL, Shah AV, Starks LT, Martin-Garrido A, Manavaki R, Yu E, Kuc RE, Grassi L, Kreuzhuber R, Kostadima MA, Frontini M, Kirkpatrick PJ, Coughlin PA, Gopalan D, Fryer TD, Buscombe JR, Groves AM, Ouwehand WH, Bennett MR, Warburton EA, Davenport AP, Rudd JH. Detection of Atherosclerotic Inflammation by 68Ga-DOTATATE PET Compared to [18F]FDG PET Imaging. J Am Coll Cardiol. 2017 Apr 11;69(14):1774-1791. doi: 10.1016/j.jacc.2017.01.060. PMID 28385306
- [Result] Corovic A, Wall C, Nus M, Gopalan D, Huang Y, Imaz M, Zulcinski M, Peverelli M, Uryga A, Lambert J, Bressan D, Maughan RT, Pericleous C, Dubash S, Jordan N, Jayne DR, Hoole SP, Calvert PA, Dean AF, Rassl D, Barwick T, Iles M, Frontini M, Hannon G, Manavaki R, Fryer TD, Aloj L, Graves MJ, Gilbert FJ, Dweck MR, Newby DE, Fayad ZA, Reynolds G, Morgan AW, Aboagye EO, Davenport AP, Jorgensen HF, Mallat Z, Bennett MR, Peters JE, Rudd JHF, Mason JC, Tarkin JM. Somatostatin Receptor PET/MR Imaging of Inflammation in Patients With Large Vessel Vasculitis and Atherosclerosis. J Am Coll Cardiol. 2023 Jan 31;81(4):336-354. doi: 10.1016/j.jacc.2022.10.034. PMID 36697134